CLINICAL TRIAL: NCT00126256
Title: Randomized Trial of Treatment Strategy for Chemotherapy in Colorectal Cancer, FFCD 2000-05
Brief Title: Trial Comparing Two Strategies of Chemotherapy for Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Collaborators: Fondation Francaise de Cancerologie Digestive (Other); Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FFCD 2000 - 05; CET 815
Record Dates: First submitted 2005-08-02; First posted 2005-08-03 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Colorectal Cancer; Metastasis
Keywords: Colorectal cancer; metastatic; chemotherapy; randomized trial
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — Fluorouracil; Leucovorin; Irinotecan; Oxaliplatin

INTERVENTIONS:
Drug: 5-fluorouracil
Drug: leucovorin
Drug: irinotecan
Drug: oxaliplatin

SUMMARY:
The standard treatment of metastatic colorectal cancer is based on systemic chemotherapy. Several effective drugs are currently available and can be administered either sequentially or in combination. Most patients receive 2 or 3 lines of chemotherapy. The aim of this randomized trial is to evaluate the potential benefit of a bitherapy with 5-fluorouracil (5-FU) and oxaliplatin as first line chemotherapy compared with a sequential chemotherapy with 5-FU alone as first line chemotherapy followed by the combination of 5-FU with oxaliplatin in case of progressive disease, in terms of progression-free survival and overall survival in patients with advanced colorectal cancer.

DETAILED DESCRIPTION:
Background:

The addition of oxaliplatin and irinotecan to 5-FU improves tumor response rate and progression-free survival in patients with advanced colorectal cancer compared with 5-FU alone, but increases toxicity. It is not clear whether such combination therapies (5-FU+oxaliplatin or 5-FU+irinotecan) should be systematically used as first line treatment or as second line treatment after 5-FU failure.

Design: open-label, multicentric, randomized trial

Aim: The main objective of this multiline strategy trial was to compare two 5-FU based regimens with or without the addition of oxaliplatin to 5-FU in the first line setting in terms of progression-free survival after two lines of chemotherapy in patients with metastatic colorectal cancer.

Treatment compared:

Control arm: first line, 2-hour infusion 400 mg/m² leucovorin (LV) followed by 5-fluorouracil 400 mg/m² and 46-hours 2,400 mg/m² every 2 weeks (LV5FU2), second line, LV5FU2 + oxaliplatin 100 mg/m² as a 2-hour perfusion on day 1 (FOLFOX6), third line, LV5FU2 + irinotecan 180 mg/m² (FOLFIRI)

Experimental arm: first line, FOLFOX6, second line, FOLFIRI, third line, 5-FU 250 mg/m²/day in continuous perfusion 7 out of 8 weeks or capecitabine 2,500 mg/m² per oral 14 out of 21 days or inclusion in a phase I

Inclusion criteria:

* Histologically confirmed metastatic colorectal adenocarcinoma
* Unresectable metastasis
* Bidimensionally measurable disease (WHO criteria)
* WHO performance status of 2 or less
* Adequate hematologic, renal function and liver functions
* No previous chemotherapy other than previous adjuvant chemotherapy or concomitant chemoradiotherapy with 5-fluorouracil and leucovorin for the treatment of the primary tumor completed at least 6 months before inclusion
* Signed written inform consent
* Quality of life questionnaire (QLQ C-30) filled out

Exclusion criteria:

* Pregnant or breast-feeding women
* No possible regular follow-up for psychological, social or geographical reason
* Severe cardiac, respiratory, renal or hepatic failure
* Active coronary heart disease
* Central nervous system metastases
* Past history of second malignancies
* Another investigational drug
* Chronic inflammatory bowel disease
* Previous chemotherapy with irinotecan or oxaliplatin based regimens

Randomization:

Randomization is performed centrally using a minimization technique, stratifying patients according to centre, previous adjuvant treatment, WHO performance status, and number of metastatic sites

Outcomes:

Progression-free survival after two lines of chemotherapy, defined as the time duration from randomization until progression after two lines of chemotherapy or death whatever the cause in the absence of progression or last-follow-up.

Overall survival, secondary surgery, response rate, progression-free survival after the first and the third line of chemotherapy, safety, quality of life and costs

Follow-up:

Tumor assessments is performed every 8 weeks, quality of live assessment every 8 weeks until progression after 2 lines of chemotherapy or for one year if no progression. After the end of the planned treatment, patients are followed up until death or the cut-off date.

Sample size and statistical analyses:

570 patients, 285 per arm will be needed to detect a difference in median of progression-free survival after two lines of chemotherapy of 3 months from 10 months in the control arm to 13 months in the experimental arm, for a type I error of 5% and a power of 80% (bilateral log rank test).

The analysis will be performed according to the intent-to treat principle. An interim analysis is planned after the inclusion of 400 patients with 3 months follow-up or the occurrence of 250 events and reviewed by an independent data monitoring committee.

Estimated duration of the trial: accrual period, 3 years, minimum follow-up, one year

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic colorectal adenocarcinoma
* Unresectable metastasis
* Bidimensionally measurable disease (World Health Organization [WHO] criteria)
* WHO performance status of 2 or less
* Adequate hematologic functions (neutrophil count, at least 1500 per cubic millimeter; and platelet count, at least 100,000 per cubic millimetre)
* Adequate renal function (serum creatinine, less than 125 micromol per liter)
* Adequate liver function (bilirubin, not more than 5 times the upper limit of normal)
* No previous chemotherapy other than previous adjuvant chemotherapy or concomitant chemoradiotherapy with 5-fluorouracil and leucovorin for the treatment of the primary tumor completed at least 6 months before inclusion
* Signed written inform consent
* Quality of life questionnaire (QLQ C-30) filled out

Exclusion Criteria:

* Pregnant or breast - feeding women
* Impossibility of regular follow-up for psychological, social or geographical reason
* Severe cardiac, respiratory, renal or hepatic failure
* Active coronary heart disease
* Patients with a history of a psychological illness or condition such as to interfere with the patient's ability to understand the requirements of the study
* Central nervous system metastases
* Past history of second malignancies
* Another investigational drug
* Chronic inflammatory bowel disease
* Previous chemotherapy with irinotecan or oxaliplatin based regimens

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 570 (Estimated)
Dates: Start 2002-02; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Progression-free survival after two lines of chemotherapy, defined as the time duration from randomization until progression after two lines of chemotherapy or death whatever the cause in the absence of progression or last-follow-up

SECONDARY OUTCOMES:
Overall survival
Secondary surgery
Response rate
Progression-free survival after the first and the third line of chemotherapy
Safety
Quality of life
Costs

CONTACTS AND LOCATIONS:
Overall Officials: Michel Ducreux, Pr, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris; Jean-Pierre F Pignon, MD, PhD, Study Director — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Institut Gustave-Roussy, Villejuif, France

REFERENCES:
- [Derived] Penichoux J, Michiels S, Bouche O, Etienne PL, Texereau P, Auby D, Rougier P, Ducreux M, Pignon JP; FFCD 2000-05 trial investigators. Taking into account successive treatment lines in the analysis of a colorectal cancer randomised trial. Eur J Cancer. 2013 May;49(8):1882-8. doi: 10.1016/j.ejca.2013.02.006. Epub 2013 Mar 13. PMID 23490654
- [Derived] Ducreux M, Malka D, Mendiboure J, Etienne PL, Texereau P, Auby D, Rougier P, Gasmi M, Castaing M, Abbas M, Michel P, Gargot D, Azzedine A, Lombard-Bohas C, Geoffroy P, Denis B, Pignon JP, Bedenne L, Bouche O; Federation Francophone de Cancerologie Digestive (FFCD) 2000-05 Collaborative Group. Sequential versus combination chemotherapy for the treatment of advanced colorectal cancer (FFCD 2000-05): an open-label, randomised, phase 3 trial. Lancet Oncol. 2011 Oct;12(11):1032-44. doi: 10.1016/S1470-2045(11)70199-1. Epub 2011 Sep 6. PMID 21903473